CLINICAL TRIAL: NCT00771836
Title: Airway Reactivity in Children Before and After Bone Marrow Transplantation
Brief Title: Airway Reactivity in Children Before and After BMT Bone Marrow Transplantation
Acronym: AHR
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: no sponsor, Rambam Medical Center, Haifa, Israel
Other Study IDs: RambamMC1866CTIL; AHRBMT1866
Record Dates: First submitted 2008-05-27; First posted 2008-10-15 (Estimated); Last update posted 2008-10-15 (Estimated); Status verified 2008-10

CONDITIONS: Cancer
Keywords: Stem cell transplantation; Airway hyper-reactivity; methacholine; pediatric
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Not retained
Oversight: Data Monitoring Committee: No

SUMMARY:
Background: Stem cell transplantation (SCT) is associated with pulmonary complications and may lead to high morbidity and mortality. We encountered several children post-SCT with a clinical picture suggestive of airway hyper-reactivity (AHR) and evidence of reversible airway obstruction that was not reported pre-transplant. Our aim was to determine if SCT induced AHR as assessed by methacholine challenge test (MCT) and to determine any correlation between AHR and pulmonary complications.

Methods: Prospective study evaluating consecutive patients referred for SCT to the Department of Pediatric Hemato-Oncology at Meyer Children's Hospital. Evaluation included pulmonary function test and methacholine challenge test before and after the transplantation, and assessment of pulmonary complications.

DETAILED DESCRIPTION:
We encountered several children post SCT with clinical picture suggestive of airway hyper-reactivity (AHR) by spirometric evidence of reversible airway obstruction that was not reported pre transplantation. Our question was if AHR is present but undiagnosed pre BMT or AHR is developed post transplantation.

Our aim was to determine if BMT induces AHR as assessed by methacholine challenge test (MCT) and to determine a possible correlation between AHR and pulmonary complications. The study was Prospective. Subjects: consecutive patients were referred for pulmonary function tests (PFT's); MCT and clincical evaluation before SCT and were followed after transplantation for at least a year. The study was approved by the ethics committee and parental consent was obtained. Clnical evaluation included medical history: type of disease, previous chemo/radiotherapy. Type of SCT was recorded (allogeneic/ autologous). respiratory evaluation included: Respiratory history; previous asthma medications; allergy/ parental smoking; Physical exam; CXR O2-Sat. on rest and exercise. PFT's included: Spirometry, lung volumes, diffusion capacity; MCT prior and 2-6 months post SCT; Follow-up: 6-12 months post SCT. Pulmonary complication: Any respiratory symptoms or signs: cough, SOB, hemoptysis, hypoxemia; New chest radiological finding; Number of hospitalizations due to pulmonary complications.

Statistics: Sample size-26 patients to detect an increase of 0.5SD in AHR with a power of 80%. No. of children with AHR before and after SCT.; Pulmonary complications and AHR: hospitalizations for pulmonary complications and AHR.

ELIGIBILITY:
Inclusion Criteria:

* age 4.5-20 years
* ability to perform spirometry consistently
* FEV1>70% predicted

Exclusion Criteria:

* FEV1<70%
* inability to perform methacholine challenge test before and after stem cell transplantation.

Ages: 4 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children who underwent SCT in the Department of Pediatric Hemato-Oncology at Meyer Children's Hospital and were referred to the Pediatric Pulmonary Unit.
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2004-07; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Positive MCT after SCT may be associated with increased risk of pulmonary complications | 3 years followup

SECONDARY OUTCOMES:
The number of patients with airway reactivity increased after after SCT (p < 0.05; McNemar test). | 3 years followup

CONTACTS AND LOCATIONS:
Overall Officials: Lea Bentur, MD, Study Director — Rambam Health Care Campus
Locations (1):
- Pediatric Pulmonary Unit, Meyer Children's Hospital of Haifa, Meyer Children's Hospital, Rambam Medical Center, and the Bruce Rappaport Faculty of Medicine, Haifa, Israel